CLINICAL TRIAL: NCT06104774
Title: Vice Superintendent
Brief Title: The Effects of a Family-Centered Tai Chi Exercise on Lung Function and Mental Health of Patients After Thoracoscopic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hsin-Yuan Fang, Vice Superintendent, China Medical University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: d17573
Record Dates: First submitted 2023-10-18; First posted 2023-10-27 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Thoracic Neoplasms
Keywords: Tai Chi exercise; Lung cancer; thoracoscopic surgery; Lung function; Mental Health; Sleep; Family-Centered
MeSH Terms: conditions — Thoracic Neoplasms; Lung Neoplasms; Psychological Well-Being | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai Chi group (Experimental): After recruitment, participants will receive Tai Chi Exercise teaching. In the acupressure group, participants will receive acupressure treatment.
  Interventions: Behavioral: Tai Chi Exercise
- Control group (No Intervention): conventional treatment

INTERVENTIONS:
Behavioral: Tai Chi Exercise — The experimental group will receive Tai Chi exercise and routine treatment after the operation, and after discharge from the hospital, they will perform Tai Chi exercise three times a week, 50 minutes each time, for a total of eight weeks after discharge.
  Arms: Tai Chi group

SUMMARY:
To explore the effect of a family-centered, eight-week, progressive sit-to-stand Tai Chi exercise on lung function and mental health in patients after thoracoscopic surgery_

DETAILED DESCRIPTION:
Lung cancer is the top death among cancers in Taiwan. The surgical excision of lung tissue is unable to regenerate new tissue after thoracoscopic lobectomy, resulting in decreased lung function and affecting health-related quality of life. 29% of female patients who received thoracic surgery tended to be anxious and depressed, and more than 60% of the family caregivers experienced mild to moderate caregiving burden and anxiety. Tai Chi exercise is a gentle exercise that can effectively enhance lung function. However, there is a lack of literature on the effects of Tai Chi exercise on lung function and mental health after thoracoscopic surgery.Methods: Exploratory sequential mixed methods study design will be used. The first phase will be a quasi-experimental study that will use purposive sampling to recruit thoracoscopic surgical patients and their family caregivers. It is estimated to enroll 60 pairs of patients and their family caregivers. The participants will be divided into experimental and control groups according to the sequential time of admission. The experimental group will receive Tai Chi exercise and routine treatment after the operation, and after discharge from the hospital, they will perform Tai Chi exercise three times a week, 50 minutes each time, for a total of eight weeks after discharge; the control group will receive conventional treatment. Repeated measures analysis of variance (repeated ANOVA) will be used for comparison between the experimental group and the control group and within the group; for other confounding factors, generalized estimating equations (GEE) will be used for analysis. In the second stage, after eight weeks of Tai Chi exercise, semi-structured interviews with about 10 patients and their caregivers will be conducted to collect their experiences and feelings related to the Tai Chi exercise. Qualitative data will be used to comprehend the quantitative data.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized to receive thoracoscopic lobectomy, wedge/partial resection, lobectomy, or sleeve resection.
2. American Society of Anesthesiologists (ASA) physiological status classification I-II (ASA, 2019).ASA Physical Status Class I: A healthy person who is healthy and does not smoke or drink.ASA physical status class II: People with mild chronic diseases but no substantial functional limitations.
3. Those who can walk on their own without any impairment in limb movement.
4. Able to communicate in Chinese or Taiwanese.

Exclusion Criteria:

1. Individuals requiring chemotherapy and radiation therapy for malignant tumors.
2. Those who have practiced Tai Chi, Qigong, external elixir exercises, or pulmonary exercises within the past year.
3. Anticipating hospitalization or surgical treatment within the next three months.
4. Individuals with musculoskeletal or peripheral vascular diseases.
5. Individuals with visual impairment, intellectual disabilities, or memory loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
vital capacity (VC) | admission day, discharge 1 day, 7 day after discharge, one month after discharge, two months after discharge
  data will be collected through lung function test
forced vital capacity (FVC) | admission day, discharge 1 day, 7 day after discharge, one month after discharge, two months after discharge
  data will be collected through lung function test
forced expiratory volume in one second (FEV1) | admission day, discharge 1 day, 7 day after discharge, one month after discharge, two months after discharge
  data will be collected through lung function test

SECONDARY OUTCOMES:
Hospital anxiety and depression scale composite | Baseline (Before operation), immediately post-operation, discharged 1 day, one week after discharge, one month after discharge, two months after discharge
  This scale measures the feelings of anxiety and stress that one has experienced in the past week. It has a total of 14 questions, including 7 questions each for the Anxiety Scale (HADS-A) and the Depression Scale (HADS-D). It is measured on a 4-point Likert scale. Score method (0-3), the total score of each item is 0-21 points, the higher the score measured by the scale, the higher the degree of anxiety and depression. The Cronbach's α coefficients of the internal consistency reliability of HADS-A and HADS-D are respectively 0.82-0.74, with high internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Hsing-Chi Hsu, Ph.D, Principal Investigator — HungKuang University, Taiwan; Kai-yu Tseng, Ph.D, Principal Investigator — Central Taiwan University of Science and Technology
Locations (1):
- China Medical University, Taichung, North Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No